CLINICAL TRIAL: NCT07288879
Title: A Multi-center Single Arm Phase II Study to Evaluate the Safety and Efficacy of Genetically Engineered Autologous Cells Expressing Anti-CD20 and Anti-CD19 Specific Chimeric Antigen Receptor in Subjects With Relapsed and/or Refractory Diffuse Large B Cell Lymphoma.
Brief Title: DALY II Japan/MB-CART2019.1 for DLBCL
Acronym: DALY II Japan
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Miltenyi Biomedicine GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M-2023-413; jRCT2033250384 (Other: Japan Registry of Clinical Trials)
Record Dates: First submitted 2025-11-20; First posted 2025-12-17 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: DLBCL - Diffuse Large B Cell Lymphoma; CAR T Cell Therapy
Keywords: CAR T Cell therapy; DLBCL
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MB-CART2019.1 in DLBCL (Experimental): MB-CART2019.1 Treatment
  Interventions: Biological: MB-CART2019.1

INTERVENTIONS:
Biological: MB-CART2019.1 — CAR T cell therapy

SUMMARY:
DALY II Japan is a phase II, multi-center, single arm study to evaluate the efficacy, safety, and pharmacokinetics of zamtocabtagene autoleucel (MB-CART2019.1) in patients with relapsed and/or refractory diffuse large B cell lymphoma (DLBCL) after receiving at least two lines of therapy.

DETAILED DESCRIPTION:
A prospective, single arm, open label, multi-center, phase II study of autologous T cells engineered against both CD19 and CD20 antigens for subjects with relapsed or refractory DLBCL after receiving at least two lines of therapy. The investigational agent is the MB-CART2019.1 cells. After successful screening, subjects will undergo leukapheresis to collect product for manufacturing. In preparation for the fresh product infusion, subjects will undergo a lymphodepleting regimen with cyclophosphamide and fludarabine. Cell infusion will be administered intravenously at a dose of 2.5 x 10^6 CAR+ cells/kg body weight. Subjects will be followed for up to 2 years, for efficacy and safety outcomes as well as health-related quality of life (HRQoL). Additional long-term follow-up will be conducted for participants under a separate long-term follow-up protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed DLBCL or associated subtype, defined by WHO 2016 classification:

   * DLBCL not otherwise specified (NOS)
   * High-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements
   * High-grade B-cell lymphoma, NOS
   * Primary mediastinal (thymic) large B-cell lymphoma
   * Transformed lymphoma (e.g. transformed follicular or marginal zone lymphoma, follicular lymphoma Grade 3B)
2. Relapsed or refractory disease after 2 or more lines of chemotherapy including rituximab and anthracycline and either having failed autologous stem cell transplant (ASCT), or being ineligible for or not consenting to ASCT 2.1 Chemotherapy-refractory disease is defined as one of the following:

   * No response to last line of therapy:

     * Progressive disease (PD) as best response to most recent therapy regimen
     * Stable disease (SD) as best response to most recent therapy with duration no longer than 6 months from last dose of therapy OR
   * Relapsed or persistent disease after prior ASCT for lymphoma

     * Disease progression or relapse less than or equal to 24 months of ASCT
     * If salvage therapy is given post-ASCT, the individual must have had no response to or relapsed after the last line of therapy 2.2 Disease relapse in subjects without prior ASCT is defined as relapse of disease in ≤ 12 months after the last dose of most recent therapy regimen 2.3 Ineligible for ASCT is defined as meeting one of the following criteria:
   * Chemotherapy-refractory disease after salvage therapy
   * Disease progression or relapse ≤ 12 months after salvage therapy
   * Intolerance to salvage therapy

   In addition, all subjects must have:
3. Age ≥18 years
4. Eastern Cooperative Oncology Group (ECOG) performance status that is either 0 or 1 at screening. ECOG performance status of 2 at screen is allowed if the decrease in performance status is due to DLBCL
5. Measurable disease according to Lugano 2014 criteria for assessing fluorodeoxyglucose-positron emission tomography (FDG-PET)/computer tomography (CT) in lymphoma (Cheson et al, 2014)
6. CD19 or CD20 antigen expression on tumor is not required after the most recent chemoimmunotherapy; however, 6.1 Subject must have at least 20 unstained slides of tissue available prior to MB-CART2019.1 infusion 6.2 If archival tissue is not available, subject must be willing to undergo attempted repeat biopsy
7. No clinical suspicion of central nervous system (CNS) lymphoma
8. If the subject has history of CNS disease, then he/she must 8.1. Have no signs or symptoms of CNS disease 8.2. Have no active disease on magnetic resonance imaging (MRI) 8.3. Have no large cell lymphoma present in cerebral spinal fluid (CSF) on cytospin preparation and flow cytometry, regardless of the number of white blood cells (WBCs)
9. If the subject has history of cerebral vascular accident (CVA) 9.1. The CVA event must be greater than 12 months prior to leukapheresis 9.2. Any neurological deficits must be stable
10. An estimated creatinine clearance by Cockcroft-Gault Equation (eGFR) > 60mL/min
11. Cardiac ejection fraction (EF) ≥ 45% as determined by an echocardiogram (ECHO)
12. Resting O2 saturation >90% on room air
13. Serum alanine aminotransferase (ALT) / aspartate aminotransferase (AST) <5 times the Upper Limit of Normal (ULN) for age
14. Total bilirubin <1.5 mg/dl, except in individuals with Gilbert's syndrome
15. Absolute neutrophil count (ANC) > 1000/μL
16. Absolute lymphocyte count > 100/μL
17. Platelet count > 50,000/μL
18. Estimated life expectancy of more than 3 months other than primary disease
19. Subjects of childbearing or child fathering potential must be willing to practice birth control from the time of enrollment on this study until the follow-up period of the study

Exclusion Criteria:

1. Primary CNS lymphoma
2. Richter's transformed DLBCL arising from chronic lymphocytic leukemia (CLL)
3. Unable to give informed consent
4. Known history of infection with human immunodeficiency virus (HIV) or active hepatitis B (HBsAg positive), unless confirmed to be polymerase chain reaction (PCR) negative; antiviral prophylaxis is required as recommended in the Japanese guidelines for Hepatitis B treatment if HBsAg negative and anti-HBc positive
5. Known history of infection with hepatitis C virus (anti-HCV positive) unless viral load is undetectable per quantitative PCR and/or nucleic acid testing
6. Known history of active seizure or presence of seizure activities or on active anti-seizure medications within the prior 12 months
7. Known history of CVA within prior 12 months
8. Known history or presence of autoimmune CNS disease, such as multiple sclerosis, optic neuritis or other immunologic or inflammatory disease
9. Presence of active CNS disorder that, in the judgment of the investigator, may impair the ability to evaluate neurotoxicity
10. Active systemic fungal, viral or bacterial infection
11. Pregnant or breast-feeding woman
12. Previous or concurrent malignancy with the following exceptions:

    * Adequately treated basal cell or squamous cell carcinoma (adequate wound healing is required prior to study entry)
    * In situ carcinoma of the cervix or breast, treated curatively and without evidence of recurrence for at least 2 years prior to the study
    * Adequately treated breast or prostate carcinoma on hormonal therapies such as Lupron or tamoxifen and in clinical remission of ≥ 2 years
    * A primary malignancy which has been completely resected / treated with curative intent and in complete remission of ≥ 2 years
13. History of non-neurologic autoimmune disease (e.g. Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus) requiring systemic immunosuppressive or systemic disease modifying agents within the last 2 years
14. Medical condition requiring prolonged use of systemic corticosteroids equivalent to Prednisone >10 mg/day
15. History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 6 months of enrollment
16. Concurrent radiotherapy (allow up to time of leukapheresis)
17. Baseline dementia that would interfere with therapy or monitoring, determined using Immune Effector Cell-Associated Encephalopathy (ICE) Assessment at baseline. (Appendix 6, Section 13.6)
18. History of severe immediate hypersensitivity reaction to any of the agents used in this study
19. Refusal to participate in additional lentiviral gene therapy LTFU protocol
20. Prior CAR T cell therapy for any indication
21. Prior allogeneic stem cell transplant for any indication.
22. Prior bispecific antibodies for cancer therapy
23. Prior T cell receptor-engineered T cell therapy
24. Prior anti CD 19 immunotherapy
25. Hypersensitivity against any drug including MB-CART2019.1 (and the constituents used in the production, ingredients/impurities, including bovine and rodent-derived components), that is scheduled or likely to be given during trial participation, e.g. as part of the mandatory preparative chemotherapy or rescue medication/salvage therapies for treatment related toxicities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 1 month
  Objective Response Rate (ORR) (complete response rate [CRR] + partial response rate [PRR]) using Lugano 2014 Criteria (Cheson et al, 2014) at one month with independent central review

SECONDARY OUTCOMES:
Complete Response Rate | 6 months
  Complete response rate using Lugano 2014 Criteria (Cheson et al, 2014) at 6 months.
Duration of response | up to 2 years
  Duration of response (DOR)
Objective Response Rate | 6 months
  ORR using Lugano 2014 criteria (Cheson et al, 2014) at 6 months.
Best Overall Response | 2 years
  Best overall response (BOR)
Progression Free Survival | up to 2 years
  Progression Free Survival
Overall Survival | up to 2 years
  Overall Survival
Type, frequency, and severity of adverse events (AEs), serious adverse events (SAEs) and adverse events of special interest (AESI) | up to 2 years
  Type, frequency, and severity of adverse events (AEs), serious adverse events (SAEs) and adverse events of special interest (AESI)
Incidence of anti-MB-CART2019.1 antibodies | up to 2 years
  Incidence of anti-MB-CART2019.1 antibodies
Persistence of MB-CART2019.1 | up to 2 years
  Persistence of MB-CART2019.1
Cytokine levels | up to 2 years
  Measure and correlate the types and level of cytokines in subjects following MB-CART2019.1 infusion with severity of CRS, ICANS and efficacy.
CD19 and CD20 antigen expression | up to 2 years
  Correlate the changes in tumor CD19 and CD20 antigen expression with disease progression and relapse
Quality of Life /Patient-Reported Outcome assessments: EQ-5D-5L Health-Related Quality of Life Index Score | Baseline, Month 3, Month 6, Month 9, Month 12, Month 18, Month 24
  Measured using the EQ-5D-5L instrument. The index score reflects health utility (range -0.281 to 1.000), where higher scores indicate better self-reported health status.
Quality of Life /Patient-Reported Outcome assessments: Functional Assessment of Cancer Therapy-Lymphoma (FACT-Lym) Total Score | Baseline, Month 3, Month 6, Month 9, Month 12, Month 18, Month 24
  The FACT-Lym is a patient-reported outcome instrument designed to assess health-related quality of life in patients with lymphoma. The total score is derived from the FACT-General core questionnaire (physical, social/family, emotional, and functional well-being) and a lymphoma-specific subscale. Higher scores indicate better health-related quality of life.

CONTACTS AND LOCATIONS:
Locations (5):
- Japan (5):
  - National Cancer Center Hospital, Tokyo
  - Toranomon Hospital, Tokyo
  - Juntendo University Hospital, Tokyo
  - Tokyo Metropolitan Komagome Hospital, Tokyo
  - Keio University Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: No